CLINICAL TRIAL: NCT04694456
Title: Pro-inflammatory Cytokines as Potential Therapeutic Target in Type 1 Facioscapulohumeral Muscular Dystrophy: Pilot Study
Brief Title: Pro-inflammatory Cytokines in Facioscapulohumeral Muscular Dystrophy (CYTOKINE-FSH)
Acronym: CYTOKINE-FSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-AOI-13
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Muscular Dystrophies
MeSH Terms: conditions — Muscular Dystrophies | interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Intervention Model Description: Interventional pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Facioscapulohumeral muscular dystrophy (Experimental): Adult ambulant patients with facioscapulohumeral muscular dystrophy type 1 (FSHD1)
  Interventions: Other: cytokines dosage; Procedure: test of walk; Procedure: Manual muscular test; Procedure: Motrice fonction mesurement

INTERVENTIONS:
Other: cytokines dosage — Mesure of cytokines concentration in serum
  Other Names: biological analysis
Procedure: test of walk — patient must walk during 6 minutes on a flat surface
Procedure: Manual muscular test — test performed to evaluate the patient muscular weakness
Procedure: Motrice fonction mesurement — scale allowing the evaluation of patient posture and upper body movements

SUMMARY:
The facial-glenohumeral muscular dystrophy type 1 (DMFSH1) is characterized by a selective and asymmetrical involvement of the facial muscles, the shoulder girdle and the anterolateral lodge legs. Genetically, the disease is transmitted in an autosomal dominant manner and is caused by a pathogen contraction of repeat units (UR) say D4Z4 localized to the telomeric portion of chromosome 4qA. The loss of UR causes hypomethylation of DNA and chromatin relaxation of the region that lead to inappropriate expression of DUX4 retrogene highly toxic. The inappropriate expression induces a T cell reaction inflammatory response that participate and increase muscle damage. In favor of this hypothesis, several muscle MRI studies have shown that atrophy and fibro-adipose degeneration (hyper signal in T1) were preceded by the appearance of muscle inflammation (hyper signal T2STIR) confirmed on histologically and dysregulation of genes involved in adaptive and innate immunity. scientific hypothesis and potential benefits: the investigateur hypothesize that in patients of DMFSH1, the immune system cells may participate in the pathophysiology of the disease through changes in serum secretion of one or more cytokines and / or a modification of the response of inflammatory cells in some cell damage stimuli. Design: this is a single-center pilot study, interventional. In this study, the investigator will assay the serum cytokines and changes in peripheral blood cells of the expression of cytokines in response to some stimuli in 20 patients with Type 1 DMFSH genetically confirmed at an intermediate stage of clinical disease (kept walking, but at least one muscle of lower limbs reached) and compare with controls from the CYTOKINAGE study. The investigator will also carry patients clinical testing (MMT sum score) and functional (6minute test march MFM) and a MRI not injected whole body (T1 sequences + and T2STIR) to study the relationship between these parameters and secretion cytokines or serum in response to certain stimuli Main objective: to compare serum levels of IL-6 in patients with DMFSH and controls.

ELIGIBILITY:
Inclusion Criteria:

* male or female age 18 to 75
* suffering from genetically confirmed FSHD1 (<11 D4Z4 repeat units on permissive chromosome 4 allele)
* ambulant or walking with assistance
* Manual Muscle Testing ≥4 for 1 of lower limb muscles

Exclusion Criteria:

* pregnancy or breast feeding
* stay in tropical/subtropical country within 3 months
* physical exercice within 10 hours
* specific diet (e.g. hypocaloric or cholesterol lowering diet)
* regular alcohol consumption; drug consumption within 3 months
* immunosuppressive or immonumodulating drug within 2 weeks or for more than 3 months withing last 6 months
* vaccination, blood transfusion of immunoglobulin treatment within 3 months
* infection within 3 weeks; HIV, HBV, HCV seropositivity
* chronic inflammatory and/or autoimmune or allergic disease from the gut (Crohn disease, ulcerative colitis), skin (psoriasis, atopic dermatitis), joints (rhumatoid arthritis), nervous system (multiple sclerosis), diabetes type I and II
* neurodegenerative disorders (Alzheimer's or Parkinson's diseases)
* diagnosed cancer not under remission for at least 5 years
* participation in the last 3 months in a research clinical trial with exposure to a pharmaceutical product or a medical device
* muscular MRI contraindication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Comparison of serum IL-6 levels between FSHD1 patients and control subjects (from other previous studies) comparable in terms of age and sex | 21 months
  Serum IL-6 levels will be measured using v-plex technology (MSD) in FSHD1 patients and compared with results obtained in paired control subjects from 2 cohorts (NCT00998231 and Cytokinage study NCT02660723)

SECONDARY OUTCOMES:
Comparison of serum levels of 28 oher pro-inflammatory cytokines between FSHD1 patients and control subjects | 21 months
  Serum levels of 28 other cytokines will be measured using v-plex technology (MSD) in FSHD1 patients and compared with results obtained in paired control subjects
Comparison of cytokines produced upon in vitro stimulation of blood cells in FSHD1 patients and control subjects | 21 months
  Cytokine production will be induced in blood cells by non-specific stimulation with LPS, ATP+LPS-EB or poly (I:C) in FSHD1 patients and compared with results obtained in control subjects
Evaluation of potential correlations between cytokines levels (either in the serum or produced upon in vitro stimulation) and clinical severity in FSHD1 patients | 21 months
  Clinical severity and muscle impairment will be evaluated using standardized clinical scales (Manual Muscle Testing, Motor Function Measure-32, 6-minute walk test, age-corrected Clinical Severity Score)
Evaluation of potential correlations between cytokines levels (either in the serum or produced upon in vitro stimulation) and muscle MRI caracteristics in FSHD1 patients | 21 months
  Whole body MRI will be recorded (T1 and T2STIR sequences) in order to evaluate muscle oedema, inflammation and degeneration

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No